CLINICAL TRIAL: NCT05059509
Title: An Open Labeled Exploratory Study to Evaluate Efficacy of FB825 in Adults With Atopic Dermatitis
Brief Title: Evaluate Efficacy of FB825 in Adults With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FB825CLIIS-04-AD
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2021-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FB825 (Experimental): One dose FB825, 5mg/kg, by 1 hour IV infusion on Day 1
  Interventions: Biological: FB825

INTERVENTIONS:
Biological: FB825 — FB825, 5mg/kg, by 1 hour IV infusion on Day 1

SUMMARY:
This is an open labeled exploratory study to evaluate efficacy of FB825 in adults with atopic dermatitis (AD). The study will be conduct at one medical center in Taiwan. Approximately 20 subjects with atopic dermatitis (AD), who meet the criteria for study entry, will be enrolled to the study. All eligible subjects will receive FB825, 5mg/kg, by 1 hour IV infusion on Day 1. Subjects will return to the study site on Days 15, 29 and 57 for the safety and efficacy evaluation. Subjects who premature withdraw from the study will have an end of study (EOS) visit within 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 20 and 65 years of age, inclusive.
2. The subject has a physician confirmed diagnosis of chronic atopic dermatitis based on 3 year history of symptoms defined by the Eichenfield revised criteria of Hannifin and Rajka and supported by positive allergen specific IgE (immunoglobulin E) at the screening visit.
3. Eczema Area and Severity Index (EASI) score 16 at the screening and baseline visits.
4. Investigator's Global Assessment (IGA) score 3 (5 point scale) at the screening and baseline visits.
5. 10 % body surface area (BSA) of AD involvement at the screening and baseline visits.
6. History of inadequate response to a stable (1 month) regimen of topical corticosteroids or calcineurin inhibitors as treatment for AD within 3 months before the screening visit. (The regimen of topical corticosteroids means medium to high potency, applied for at least 28 days or for the maximum duration recommended by product prescribing information.)
7. Patients must be applying stable doses of emollient provided for atopic dermatitis twice daily for at least 7 days before the baseline visit.
8. Female subjects of childbearing potential must use at least two forms of birth control. One must be barrier protection (i.e., condom or female condom) and the other is one of acceptable method of birth control (ie, diaphragm, intrauterine device, hormonal contraceptives, or abstinence) throughout the study. Subjects who are surgically sterile (ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), or postmenopausal (defined as amenorrhea for 12 consecutive months and documented serum follicle stimulating hormone level >40 mU/mL) will be considered as no childbearing potential. All female subjects must have a negative serum pregnancy test prior to dosing.

   Note: The subject must use the method of contraception mentioned above during study period and in 16 weeks or 5 half lives after the last dosing of FB825.
9. The subject has a body weight ≥ 40 kg at screening and a body mass index of 18.0 to 30.0 kg/m2, inclusive.
10. The subject has a normal, as determined by the investigator, 12 lead electrocardiogram (ECG) with normal cardiac conduction parameters:

    * Heart rate between 45 and 100 bpm;
    * Fridericia corrected QT interval (QTcF) ≤450 milliseconds (men) or ≤470 milliseconds (women);
    * QRS interval lower than 120 milliseconds.
11. The subject is healthy, except atopic diseases, as determined by the investigator, on the basis of clinical laboratory test results performed at screening. If the results are outside the normal reference ranges, the subject may be included only if the investigator judges the abnormalities or deviations from normal not to be clinically significant.
12. The subject is able to provide written informed consent.
13. The subject agrees to comply with all protocol requirements.

Exclusion Criteria:

1. Female subjects who are pregnant or lactating.
2. The subject is on diet or with poor intake.
3. The subject has a history of heart arrhythmias (any clinically relevant).
4. The subject has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody,or human immunodeficiency virus antibodies at screening.
5. The subject has a history of alcohol or drug abuse that would impair or risk the patients' full participation in the study, in the opinion of the investigator.
6. The subject is under judicial supervision or curatorship.
7. The subject has a clinically relevant, currently active or underlying gastrointestinal, cardiovascular, nervous system, psychiatric, metabolic, renal, hepatic, respiratory (with the exception of uncomplicated allergic rhinitis), inflammatory, immunological, endocrine, diabetes, or infectious disease and ineligible to participate in the study judged by investigator.
8. The subject has any history of a previous anaphylactic reaction.
9. The subject has any condition that, in the opinion of the investigator, would compromise the study or the well being of the subject or prevent the subject from meeting or performing study requirements.
10. The subject has received any immunoglobulin products or blood products within 3 months prior to dosing.
11. The subject has received an biologic product:

    * The subject has received any cell depleting agents, not only limited to rituximab, within 6 months prior to dosing, or before the lymphocyte count returns to normal, whichever is longer.
    * The subject has received other biologics within 5 half lives (if known) or 16 weeks, which is longer, prior to dosing).
12. The subject has one or more of the following laboratory abnormalities at screening as defined by Division of Microbiology and Infectious Diseases Adult Toxicity Table 2007:

    * Aspartate aminotransferase or alanine aminotransferase (>2 × upper limit of normal [ULN]) or higher
    * Total bilirubin ≥1.5 × ULN
    * Serum creatinine ≥1.6 × ULN
    * Any other laboratory abnormality higher than or equal to grade 2 with the exception of IgE level, eosinophil counts, eosinophil cationic protein (ECP) and laboratory values mentioned above.

    Note: Laboratory values may be converted to equivalent standard units. Retesting of abnormal laboratory values that may lead to exclusion will be allowed once (without prior sponsor approval). Retesting will take place during an unscheduled visit in the screening phase (before baseline).
13. The subject has received any approved or unapproved (ie, investigational) immunotherapy treatment within the past 3 months.
14. The subject has used any of the following classes of medication (prescription or over the counter):

    * Intranasal corticosteroid (eg, fluticasone propionate) within 30 days prior to dosing.
    * Systemic corticosteroids (eg, prednisone) within 30 days prior to dosing.
    * Leukotriene modifiers (eg, montelukast) within 30 days prior to dosing.
    * Immunosuppressants (eg, gold salts, methotrexate, azathioprine, cyclosporine) within the past 30 days prior to dosing.
    * Immunomodulating drugs (eg, interferon-gamma ) within the past 30 days prior to dosing.
    * Anti IgE (eg, omalizumab) within the past 1 years prior to dosing
    * Allergen immunotherapy within the past 1 years prior to dosing
    * Orally inhaled corticosteroids (eg, budesonide) within the past 30 days prior to dosing
15. The subject has received phototherapy within 4 weeks prior to dosing.
16. The subject has received live vaccine within 12 weeks prior to dosing.
17. The subject has known or suspected history of immunosuppression, including history of opportunistic infections (eg, TB) per investigator judgment.
18. The subject has history of malignancy within 5 years before the screening period.
19. High risk of parasite infection.

    * Risk factors for parasitic disease (living in an endemic area, chronic gastrointestinal symptoms, travel within the last 6 months to regions where geohelminthic infections are endemic, and/or chronic immunosuppression) AND
    * Evidence of parasitic colonization or infection on stool evaluation for ova and parasites.

Note: stool ova and parasite evaluation will only be conducted in patients with risk factors and an eosinophil count more than twice the upper limit of normal

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
The mean change in mIgE (Membrane bound Immunoglobulin E) B cell count (absolute and percentage) from baseline | week 2 and 4

SECONDARY OUTCOMES:
The mean percentage change in Pruritus Visual Analogue Scale (VAS) from baseline | week 2 and 4
The mean percentage change in Eczema Area and Severity Index (EASI) from baseline | week 2 and 4
The mean percentage change in Severity Scoring of Atopic Dermatitis Index (SCORAD) from baseline | week 2 and 4
The mean percentage change in Investigator Global Assessment (IGA) from baseline | Weeks 2 and 4
The mean percentage change in Body Surface Area (BSA) involved in atopic dermatitis from baseline to | Weeks 2 and 4
The mean change in Dermatology Life Quality Index (DLQI) from baseline | Weeks 2 and 4

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No